CLINICAL TRIAL: NCT06069973
Title: Machine Learning and Biomarkers for Early Detection of Delayed Cerebral Ischemia
Brief Title: Using Machine Learning and Biomarkers for Early Detection of Delayed Cerebral Ischemia
Acronym: CIDAIBASSAH
Status: Recruiting | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Linda Block, Dr, Sahlgrenska University Hospital
Other Study IDs: CIDAI-BAS-SAH
Record Dates: First submitted 2023-09-26; First posted 2023-10-06 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Ischemic Stroke; Hemorrhagic Stroke
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Cerebrospinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Delayed cerebral ischemia: Definition by Vergouwen et al. Verified by computed tomography
  Interventions: Other: No intervention, observational study
- Non-delayed cerebral ischemia: No signs of cerebral ischemia clinically or by computed tomography.
  Interventions: Other: No intervention, observational study

INTERVENTIONS:
Other: No intervention, observational study — No intervention

SUMMARY:
The overall goal of this project is to determine if machine learning and analysis of neurospecific biomarkers can enable early detection of upcoming or ongoing cerebral ischaemia in patients suffering from subarachnoid haemorrhage with altered consciousness due to cerebral injury or sedation. Analyses of heart rate variability, electroencephalgraphy,nearinfrared spectroscopy, cerebral autoregulation, and brain injury specific biomarkers in blood and cerebrospinal fluid will be performed.

DETAILED DESCRIPTION:
A new and promising approach to detect ongoing cerebral ischemia might be the detection of neurospecific biomarkers in blood. A biomarker for cerebral ischaemia, similar to troponin T and troponin I for detecting cardiac ischaemia, would be precious; however, such a biomarker for cerebral ischaemia is currently lacking. (9) There are several interesting neurospecific biomarkers for this purpose, such as Glial fibrillary acidic protein (GFAP), neuron-specific enolase (NSE), total tau, S-100, and neurofilament light chains (NFL). At this point, we do not have enough knowledge about levels of neurospecific biomarkers in blood and cerebrospinal fluid during delayed cerebral ischemia after subarachnoid hemorrhage. The sampling of neurospecific biomarkers have a dual purpose, the first is to investigate if we can detect ongoing cerebral ischemia with these biomarkers, and the second purpose is to compare levels of biomarkers to outcome in mortality and morbidity determined by the Glasgow Coma Scale Extended at 1-year, 3-years and 5-years after admission.

Machine learning algorithms for predicting outcomes after delayed cerebral ischemia using a combination of clinical and imaging data have emerged. Nevertheless, prediction of delayed cerebral ischemia does not prevent it; to prevent delayed cerebral ischemia, an easily applied, cheap and reliable monitoring system that can warn physicians of the imminent risk of cerebral ischemia needs to be developed, making it possible to intervene.

The overall goal of this project is to develop methods that enable the detection of upcoming or ongoing cerebral ischaemia in patients with subarachnoid haemorrhage

Our primary aims are:

* To develop a machine learning-based model that can identify patterns in signals obtained from HRV, NIRS, and EEG monitoring, which are consistent with upcoming cerebral ischemia and provide a warning about this to attending physicians.
* To define the specificity and time relation of neurospecific biomarkers in blood and cerebrospinal fluid in patients with subarachnoid haemorrhage with and without delayed cerebral ischemia to evaluate if any of these biomarkers can be used as an indicator for ongoing cerebral ischemia.
* To assess the prognostic value of changes in physiological and neurospecific biomarkers changes during the acute phase after subarachnoid hemorrhage on long-term outcome.

ELIGIBILITY:
Inclusion Criteria:

Patients over the age of 18 with aneurysmal subarachnoid hemorrhage admitted to intensive care units at Sahlgrenska University hospital.

Exclusion Criteria:

* Unable to consent,
* Cardiac arrythmia,
* Previous brain damage

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult people with aneurysmal subarachnoid hemorrhage
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2033-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Early warning system | 2023-2033
  To develop a machine learning-based model that can identify patterns in signals obtained from HRV, NIRS, and EEG monitoring, which are consistent with upcoming cerebral ischemia and provide a warning about this to attending physicians.
  To define the specificity and time relation of neurospecific biomarkers in blood and cerebrospinal fluid in patients with subarachnoid haemorrhage with and without delayed cerebral ischemia to evaluate if any of these biomarkers can be used as an indicator for ongoing cerebral ischemia.
  To assess the prognostic value of changes in physiological and neurospecific biomarkers changes during the acute phase after subarachnoid hemorrhage on long-term outcome.
Autoregulation | 2023-2033
  xyz

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No